CLINICAL TRIAL: NCT07253064
Title: A Monocentre, Randomized, Contralateral Trial to Study the Effect of Temporal Changes in Ocular Biometry of Two Myopia Control Lenses
Brief Title: Study Comparing Eye Growth Over Time in Children Using Two Myopia Control Lenses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Essilor International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WS10449
Record Dates: First submitted 2025-09-29; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Myopia
Keywords: myopia control; axial length; choroidal thickness
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OD: MCL 1; OS: MCL 2 (Experimental): Each participant wears the study eyeglasses containing both Myopia Control Lens 1 (MCL 1) and Myopia Control Lens 2 (MCL 2) design, with one type of lens in each eye throughout the study period. For Arm 1, MCL 1 will be worn in the right eye, and MCL 2 in the left eye for a period of 6 months.
  Interventions: Device: MCL 1; Device: MCL 2
- OD: MCL 2; OS: MCL 1 (Experimental): Each participant wears the study eyeglasses containing both Myopia Control Lens 1 (MCL 1) and Myopia Control Lens 2 (MCL 2) design, with one type of lens in each eye throughout the study period. For Arm 2, MCL 2 will be worn in the right eye, and MCL 1 in the left eye for a period of 6 months.
  Interventions: Device: MCL 1; Device: MCL 2

INTERVENTIONS:
Device: MCL 1 — Myopia Control Lens 1 (MCL 1) is an ophthalmic lens intended to slow down eye growth in children. This lens will be dispensed to either the right or left eye and will be worn by the participant for a period of 6 months.
Device: MCL 2 — Myopia Control Lens 2 (MCL 2) is an ophthalmic lens intended to slow down eye growth in children. This lens will be dispensed to either the right or left eye and will be worn by the participant for a period of 6 months.

SUMMARY:
The goal of this clinical trial is to investigate the short-term changes in the eye structure while wearing two types of lenslet-based myopia control lenses over a period of 6 months in children aged 6 to 13 years with myopia. The main question it aims to answer is:

* How the eye responds, at each timepoint, to the two myopia control lenses by evaluating:

  1. Change in axial length
  2. Change in choroidal thickness

     Participants will:
* Wear the study spectacles
* Visit Essilor R&D Centre for follow-up sessions

ELIGIBILITY:
Inclusion Criteria:

* Volunteer participant
* Informed consent of parent or guardian and assent of participant
* Age: Equal to or greater than 6 years but not older than 13 years at the time of informed consent and assent.
* Refractive error (manifest refraction):

  * Equal or less than -0.50 D or equal or greater than -4.75D.
  * Astigmatism should be less than or equal to 2.00D.
* Anisometropia should be less than or equal to 1.00D
* Best corrected visual acuity: Better than 0.2 logMAR in each eye
* Willingness and ability to:

  * participate in trial for at least 6 months.
  * attend scheduled visits.
  * not to be involved in other myopia control treatments concurrently.
* No history of any myopia control interventions (i.e., myopia control spectacle lenses, myopia control contact lenses, orthokeratology lenses or atropine, etc.)

Exclusion Criteria:

* History or presence of:

  * An ocular disease
  * Strabismus
  * Amblyopia
* Currently or previously on any myopia control interventions (i.e., myopia control spectacle lenses, myopia control contact lenses, orthokeratology lenses or atropine, etc.)

Ages: 6 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-11-11 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Axial Length | Baseline, 1 hour post-dispense, 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, and 24 weeks post-dispense.

SECONDARY OUTCOMES:
Change in Choroidal Thickness | Baseline, 1 hour post-dispense, 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, 10 weeks, 12 weeks, and 24 weeks post-dispense.

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Gopalakrishnan, Principal Investigator — Essilor R&D Centre Singapore
Locations (1):
- Essilor R&D Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li X, Huang Y, Liu C, Chang X, Cui Z, Yang Q, Drobe B, Bullimore MA, Chen H, Bao J. Myopia control efficacy of spectacle lenses with highly aspherical lenslets: results of a 5-year follow-up study. Eye Vis (Lond). 2025 Mar 5;12(1):10. doi: 10.1186/s40662-025-00427-3. PMID 40038807
- [Background] Lau JK, Wan K, Cheung SW, Vincent SJ, Cho P. Weekly Changes in Axial Length and Choroidal Thickness in Children During and Following Orthokeratology Treatment With Different Compression Factors. Transl Vis Sci Technol. 2019 Jul 23;8(4):9. doi: 10.1167/tvst.8.4.9. eCollection 2019 Jul. PMID 31360614